CLINICAL TRIAL: NCT04431128
Title: Adenoid Hypertrophy, Etiology, Clinical Manifestations and Related Morbidity, Correlation With Infant Feeding Position
Brief Title: Adenoid Hypertrophy, Respiratory Complications and Correlation With Infant Feeding Position
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Avital Avraham, Prof., Hadassah Medical Organization
Other Study IDs: Clalit HS
Record Dates: First submitted 2020-06-07; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Adenoid Hypertrophy
Keywords: Adenoid hypertrophy; Allergy; Infant Feeding Position; GER; Pneumonia; Bronchitis; Otitis
MeSH Terms: conditions — Hypersensitivity; Pneumonia; Bronchitis; Otitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- study group: Adenoid hypertrophy
  Interventions: Behavioral: infant feeding position
- Control group: UTI, GE, vomiting, diarrhea
  Interventions: Behavioral: infant feeding position

INTERVENTIONS:
Behavioral: infant feeding position — correlation with allergy, GER or feeding position

SUMMARY:
500 children aged 0-5 years followed since birth by Principal Investigator (PI)since January1, 2003 till December 31, 2018 and diagnosed with adenoid hypertrophy (AH) (study group) and 500 children aged 0-5 years followed by principal investigator during the same years and diagnosed as urinary tract infection (UTI), gastroenteritis (GE), diarrhea, vomiting but without AH (control group) were compared. Morbidity and treatment will be compared and correlated with gastro-esophageal reflux (GER), allergy and infant feeding position during the first few years of life in the two groups.

DETAILED DESCRIPTION:
The 2 groups are children aged 0-5 years and treated by PI and followed since birth during years 2003-2018. Study group consists of children diagnosed at least 2 times as AH and control group as similar children with UTI, GE, vomiting or diarrhea. Respiratory problems (pneumonia, bronchopneumonia, bronchitis), ear problems (otitis media OM, serous OM), antibiotic treatment, use of bronchodilators, inhaled corticosteroid (ICS), chest X-rays, anomalous laboratory results, emergency room visits and hospitalization rates will be compared in the two groups, together with details concerning feeding position during the first years of life. Correlation between morbidity, degree of nasopharyngeal obstruction, allergy, GER and supine feeding position, will be evaluated.

ELIGIBILITY:
Inclusion Criteria: Study group: Young children with diagnosis of adenoid hypertrophy followed by PI Control group: young children with diagnosis of UTI, GE, vomiting or diarrhea followed by PI

Exclusion Criteria: Children with cystic fibrosis, primary dyskinesia, immune deficiency, congenital anatomical malformations of nasal or airway passages.

Children older than 6 months of age when starting to be followed by PI.

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Young infants followed since birth or from the first half of the first year of life, followed at least for 5 years by PI, study group (till 500 children) with the diagnosis of AH, control group (till 500 children) diagnosed as UTI, GE, vomiting or diarrhea and without AH.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-06-06 (Actual)

PRIMARY OUTCOMES:
Respiratory complications | 3 years
  Number of participants with Pneumonia, bronchitis
Ear complications | 3 years
  Number of participants with otitis media, serous otitis media

SECONDARY OUTCOMES:
Correlations between morbidity, degree of adenoid hypertrophy and feeding position | 5 years
  Correlation between respiratory morbidity, ear morbidity, laboratory and chest & nasopharynx X-rays with feeding position in first year of life
  Correlation between respiratory and ENT morbidity with degree of adenoid obstruction, allergy, GER and infant feeding position during the first 2 years of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tully SB, Bar-Haim Y, Bradley RL. Abnormal tympanography after supine bottle feeding. J Pediatr. 1995 Jun;126(6):S105-11. doi: 10.1016/s0022-3476(95)90249-x. PMID 7776069
- [Result] Konno A, Hoshino T, Togawa K. Influence of upper airway obstruction by enlarged tonsils and adenoids upon recurrent infection of the lower airway in childhood. Laryngoscope. 1980 Oct;90(10 Pt 1):1709-16. PMID 7421381
- [Result] Avital A, Donchin M, Springer C, Cohen S, Danino E. Feeding young infants with their head in upright position reduces respiratory and ear morbidity. Sci Rep. 2018 Apr 26;8(1):6588. doi: 10.1038/s41598-018-24636-0. PMID 29700412